CLINICAL TRIAL: NCT03941132
Title: Clinical Phase II/III Trial of Ustekinumab to Treat Type 1 Diabetes (UST1D2)
Acronym: UST1D2
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Janssen, LP (Industry)
Responsible Party: Principal Investigator, Jan Dutz, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H19-00411
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1D; Ustekinumab; new-onset; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Ustekinumab; Saline Solution

STUDY DESIGN:
Intervention Model Description: There will be a total of 60 patients enrolled in the study. The study participants will be enrolled at 2 centers (Vancouver and Toronto), and will be referred by adult or pediatric endocrinologists. This sample size estimation is based on results from week 52 C-peptide AUC values observed in the pilot UST1D study and the expected 1-year C-peptide decline in adult-onset T1D patients. Using a 2:1 Ustekinumab vs. placebo randomized assignment, a sample size of 60 yields 85% power to detect improvement in C-peptide function (alpha = 0.05) in the Ustekinumab group for an unstratified analysis at 12 months. Sixty-six participants (44 active: 22 placebo) will be recruited to allow for an approximate 10% loss to follow-up.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ustekinumab (Experimental): Week 0: Loading dose of 6mg/kg Ustekinumab Intravenously.
  Weeks 8, 16, 24, 32, 40, and 48 (6 visits): 90mg Ustekinumab subcutaneously.
  Weeks 28, 52, 78: Non-dosing visits where a Mixed Meal Tolerance Test will be administered.
  Total of 11 visits
  Interventions: Drug: Ustekinumab
- Saline Solution - Placebo (Placebo Comparator): Patients allocated to receive placebo will receive respective amounts of a saline-placebo at the same intervals.
  Week 0: Loading dose of 6mg/kg saline intravenously.
  Weeks 8, 16, 24, 32, 40, and 48 (6 visits): 90mg saline subcutaneously.
  Weeks 28, 52, 78: Non-dosing visits where a Mixed Meal Tolerance Test will be administered.
  Total of 11 visits
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ustekinumab — Week 0: Loading dose of 6mg/kg Ustekinumab Intravenously.
  Weeks 8, 16, 24, 32, 40, and 48 (6 visits): 90mg Ustekinumab subcutaneously.
  Other Names: Stelara
  Arms: Ustekinumab
Drug: Placebo — Patients allocated to receive placebo will receive respective amounts of a saline-placebo at the same intervals.
  Week 0: Loading dose of 6mg/kg saline intravenously.
  Weeks 8, 16, 24, 32, 40, and 48 (6 visits): 90mg saline subcutaneously.
  Other Names: Saline solution
  Arms: Saline Solution - Placebo

SUMMARY:
In type 1 diabetes (T1D), immune defense cells in the body attack and destroy insulin-producing beta cells leaving affected people with a lifelong need for daily insulin injections. Even with insulin injections, blood glucose (sugar) control is imperfect and leads to many health complications and a shortened life span. Our pilot study (NCT02117765) has informed us that Ustekinumab is safe in the treatment of participants with recent-onset T1D. Ustekinumab is currently licensed for use in psoriasis where it has proven to be both highly effective and safe. The investigators hope that if the drug can block immune cells soon after the development of diabetes, any remaining insulin-producing cells may be protected, and regenerate, thus producing more insulin so that individuals may be insulin free, or require less insulin. This trial will assess the efficacy of Ustekinumab in decreasing C-peptide decline (proxy for endogenous insulin production) in participants with recent onset T1D.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blinded, multi-centre phase II/II study to assess efficacy and safety of Ustekinumab (STELARA®) in patients with T1D. The investigators will perform a phase II/III clinical trial with a total of 66 adult (18-35 years old) subjects with recent-onset T1D. There will be two study cohorts, with a drug:placebo ratio of 2:1. Patients receiving the study drug will receive a loading dose of 6mg/kg Ustekinumab IV given at week 0. Thereafter, 90mg Ustekinumab subcutaneously given at weeks 8, 16, 24, 32, 40, 48 (total of 7 doses). Patients randomized to receive placebo will receive respective amounts of a saline-placebo. An additional non-dosing visit at the midpoint (week 28) is required to measure 2-hour C-peptide during a MMTT. Patients will be followed for 78 weeks following the first dose. There will be a total of 10 study visits over 78 weeks, three of which are non-dosing and follow-up visits. Recruitment and screening for the study will be completed within the first 24 months. The follow up period is 1 and 1.5 years from the first dose.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of type 1 diabetes mellitus in accordance with the ADA/CDA criteria.
2. An interval of ≤100 days between the diagnosis and the first dose of the study drug.
3. Ability to provide documented informed consent.
4. Male or female, aged 18-35 years inclusive, at the time of the anticipated first dose of the study drug.
5. Evidence of residual functioning β cells. This will be assessed by a C-peptide level over 0.2nmol/L in the MMTT test.
6. Positive for at least one diabetes-related autoantibody.
7. Willing to record all insulin taken and blood glucose levels that are required for monitoring during the study, including reporting any hypoglycaemic events.

Exclusion Criteria:

1. No condition that, in the investigators' judgment, is likely to cause the subject to not be able to understand information in order to provide informed consent.
2. History of malignancy.
3. No significant and/or active disease in any body system that is likely to increase the risk to the subject or interfere with the subject's participation in the study.
4. No significant systemic infection during the 6 weeks before the first dose of the study drug.
5. No history of current or past active tuberculosis infection and no latent tuberculosis as per CDC guidelines.
6. Have used any other investigational drug within the 3 months prior to the first dose and/or intend on using any investigational drug for the duration of the study.
7. Prior or current treatment that is known to cause a significant, ongoing change in the course of T1D or immunological status.
8. Current or prior (within 30 days prior to first study drug dose) use of medications known to influence glucose tolerance.
9. No significant abnormal laboratory values during the screening period, other than those due to T1D.
10. Not pregnant, breastfeeding or planning to become pregnant during the 60 days after the last dose of the study drug.
11. Have not received any live vaccines within 30 days prior to the first study drug dose and are not expected to need to receive a vaccine during the study.
12. No prior allergic reaction, including anaphylaxis, to any component of the study drug product.
13. No prior allergic reaction, including anaphylaxis, to any human, humanized, chimeric or rodent antibody treatment.
14. Have not undergone any major surgery within the 30 day period prior to the first drug dose and not anticipating requiring surgery during the study period.
15. Negative results for Hepatitis B surface antigen and for antibodies to Hepatitis B core antigen, or evidence of Hepatitis B surface antibody > 10 IU, and negative for Hepatitis C. Negative results for HIV and not considered by the investigator to be at high risk for HIV infection.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Baseline change in 2-hour mixed meal-stimulated C-peptide AUC at week 52. | Week 52
Rate, frequency and severity of all adverse events including; hypoglycemic episodes; injection reactions; hypersensitivity reactions; evidence of infection and posterior leukoencephalopathy syndrome. | Week 52

SECONDARY OUTCOMES:
2-hour MMTT-stimulated C-peptide AUC at weeks 28 and 78) | Weeks 28 and 78
HbA1C and insulin use in units per kg body weight per day at weeks 0, 8, 16, 24, 28, 32, 40, 48, 52, 78. | 78 Weeks
Immune phenotyping via flow cytometry of all IL-12, IL-23, IL-17, IFN-γ secreting immune subsets at weeks 0, 32, 52, 78). | 78 Weeks
Basic immune phenotyping of WBC subsets | 78 Weeks
HLA- A, B, C, DR, DP, DQ typing at weeks 0, 8 ,16, 32, 52, 78) | 78 Weeks
Fluorospot (ELISpot) analysis for IL-17 and IFN-γ secretion in response to whole insulin and antigens for CD8+ and CD4+ T cells. | 78 Weeks
Luminex/Mesoscale assessment of serum cytokines IL-17, IFN-γ, IL-12p40, IL-12p70 and IL-23. | 78 Weeks
Regulatory T cell (CD4+ FOXP3+): Effector T cell (CD4+ FOXP3-CD25+) ratio. | 78 Weeks
CD154 and CD134 (OX40) based assays to determine diabetogenic antigen specific responses of T helper cells. | 52 Weeks
Nanostring assessment of whole blood and PBMC RNA gene expression of IL-17 and IFN-γ family genes. | 78 Weeks
Epigenetic assessment of Treg phenotype and function. | 78 Weeks
Sequencing and profiling of microbiome. | 78 Weeks
Glycaemic variability in continuous glucose monitoring and hypoglycaemia rates. | 78 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jan Dutz, MD FRCPC, Principal Investigator — University of British Columbia; Betina F Rasmussen, MSc, Study Director — University of British Columbia
Locations (2):
- Canada (2):
  - Mount Sinai Hospital/UHN, Toronto, British Columbia
  - BCDiabetes, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Undecided